CLINICAL TRIAL: NCT03724591
Title: A Randomized Controlled Clinical Trial to Investigate the Effects of Total Mesorectum Excision With Left Colic Artery Preservation for the Treatment of Rectal Cancer
Brief Title: Total Mesorectum Excision With Left Colic Artery Preservation for the Treatment of Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRSYM201810
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Rectal Cancer
Keywords: left colic artery; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a high ligation of IMA (Experimental): total mesorectal excision (TME) for rectal cancer by a high ligation of IMA without preservation of left colic artery
  Interventions: Procedure: a high ligation of IMA
- a low ligation of IMA (Active Comparator): total mesorectal excision (TME) for rectal cancer by a low ligation of IMA with preservation of left colic artery
  Interventions: Procedure: a low ligation of IMA

INTERVENTIONS:
Procedure: a high ligation of IMA — total mesorectal excision (TME) for rectal cancer by a high ligation of IMA without preservation of left colic artery
  Arms: a high ligation of IMA
Procedure: a low ligation of IMA — total mesorectal excision (TME) for rectal cancer by a low ligation of IMA with preservation of left colic artery
  Arms: a low ligation of IMA

SUMMARY:
A randomized controlled clinical trial to compare the short and long term outcomes of left colic artery preservation for the treatment of Rectal Cancer

DETAILED DESCRIPTION:
Rectal cancer is one of most frequently diagnosed cancers and one of the leading causes of cancer death around the world. Surgery remains the main treatment for rectal cancer. Anastomosis leakage (AL) is an unresolved, devastating and lethal complication after rectal cancer surgery and remains to be a serious difficulty for surgeons despite its causes, preventions and treatments having been extensively studied.

To achieve a radical dissection of lymph nodes, it is necessary to remove the central lymph nodes at the root of inferior mesenteric artery(IMA) trunk.From the perspectives of lymph nodes dissection and tension-free anastomosis, it is preferred to perform a high ligation of IMA. However, there is still a controversy whether IMA should be high ligated or not. The argument mainly focuses on whether this performance will compromise the blood perfusion of the proximal limb of the anastomosis leading to the occurrence of AL. Some studies suggested that a high ligation did not increase the rate of AL. There are still many surgeons prefer the transection of IMA distal to the left colic artery(LCA) with the intention to preserve a good blood supply of the left colon after the performance of lymph node dissection around IMA. Some studies suggests that the preservation of LCA in anterior resection for mid and low rectal cancer is associated with lower rates of AL. Further investigations are needed to resolve the controversy.

In this study, eligible patients will be randomly allocated to receive total mesorectal excision (TME) for rectal cancer either by a high ligation of IMA without preservation of left colic artery or a low ligation of IMA with preservation of left colic artery. Postoperative complications, including anastomosis leakage, anastomosis bleeding, will be recorded. Patients will be followed up every 3 months for 2 year, every 6 months for 3 years postoperatively to study the long term effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for curative surgery over 18 years old;
* American Society of Anesthesiologists(ASA) grade I-III;
* Pathological diagnosis of rectal adenocarcinoma;
* Patients suitable for abdominalperineal resection
* Informed consent;
* No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.

Exclusion Criteria:

* Pregnant patient;
* History of psychiatric disease;
* Use of systemic steroids;
* Simultaneous multiple primary colorectal cancer;
* Preoperative imaging examination results show:1. Tumor involves the surrounding organs and combined organ resection need to be done;2. distant metastasis;3. unable to perform R0 resection;
* History of any other malignant tumor in recent 5 years;
* Patients need emergency operation: mechanic ileus, perforation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Anastomosis leakage rate | 30 days

SECONDARY OUTCOMES:
Anastomosis bleeding rate | 30 days
disease-free survival | 5 years
local recurrence rate | 5 years
operative time | 1 day
number of lymph nodes retrieved | 1 day
postoperative quality of life as assessed by EORTC QLQ-C30 questionnaire | 5 years
  Compare the differences in postoperative quality of life of patients treated with these two regimens using EORTC QLQC30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yueming Sun, PhD, Study Director — The First Affiliated Hospital with Nanjing Medical University